CLINICAL TRIAL: NCT04176393
Title: A Phase 1, Multicenter, Single-Arm Study Evaluating Pharmacokinetic, Pharmacodynamic, Safety, and Clinical Efficacy of Orally Administered Ivosidenib in Chinese Subjects With Relapsed or Refractory Acute Myeloid Leukemia With an IDH1 Mutation
Brief Title: A China Bridging Study of Ivosidenib in r/r AML Subjects With an IDH1 Mutation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS3010-101
Record Dates: First submitted 2019-10-29; First posted 2019-11-25 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ivosidenib (CS3010) tablet (Experimental): Ivosidenib (CS3010) tablet
  Interventions: Drug: ivosidenib

INTERVENTIONS:
Drug: ivosidenib — subjects will receive a single dose of ivosidenib 500 mg on Day -3 (i.e., 3 days prior to the start of daily dosing) and undergo PK/PD assessments over 72 hours to evaluate drug concentrations and 2-HG levels. Following that, subjects will be treated with ivosidenib 500 mg once a day (QD) PO continuously (28-day cycles, there are no inter-cycle rest periods).
  Other Names: TIBSOVO

SUMMARY:
This is a phase 1, multi-center, single-arm study to evaluate the pharmacokinetics(PK)/ pharmacodynamics(PD), safety, and clinical efficacy of orally administered Ivosidenib in Chinese subjects with R/R AML with an IDH1 mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be ≥ 18 years of age.
2. Subjects must have R/R AML
3. Subjects must have documented IDH1 R132 gene-mutated based on the central evaluation.
4. Subjects must have ECOG PS of 0 to 2.
5. Subjects must be amenable to serial bone marrow sampling and peripheral blood samplings during the study.
6. Subjects must have adequate hepatic function as evidenced by Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), unless considered due to Gilbert's disease or leukemic involvement and Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3.0 × ULN, unless considered due to leukemic involvement.
7. Subjects must have an adequate renal function as evidenced by Serum creatinine ≤ 2.0 × ULN or Creatinine clearance >40 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR) estimation.
8. Subjects must be recovered from any clinically relevant toxic effects of any prior surgery, radiotherapy, or other therapy intended for the treatment of cancer.

Exclusion Criteria:

1. Subjects who previously received prior treatment with a mutant-specific IDH1 inhibitor and progressed on therapy.
2. Subjects who have undergone HSCT within 60 days of the first dose of ivosidenib, or subjects on immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD).
3. Subjects who received systemic anticancer therapy or radiotherapy < 14 days prior to their first day of ivosidenib administration. Hydroxyurea and leukapheresis are allowed prior to enrollment and after the start of ivosidenib for the control of leukocytosis to reduce peripheral leukemic blasts.
4. Subjects who received an investigational agent < 14 days prior to their first day of study drug administration.
5. Subjects who received traditional Chinese medicine with known anti-cancer indication < 14 days prior to their first day of study drug administration.
6. Subjects for whom potentially curative anticancer therapy is available.
7. Subjects with an active severe infection that required anti-infective therapy or with an unexplained fever > 38.5°C during screening visits or on their first day of study drug administration (at the discretion of the Investigator, subjects with tumor fever may be enrolled).7. Subjects who are pregnant or breastfeeding.
8. Subjects with New York Heart Association (NYHA) Class III or IV congestive heart failure or LVEF < 40% by an echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within approximately 28 days of C1D1.
9. Subjects with a history of myocardial infarction within the last 6 months of screening.
10. Subjects with known unstable or uncontrolled angina pectoris.
11. Subjects with a known history of severe and/or uncontrolled ventricular arrhythmias.
12. Subjects with known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
13. Subjects with clinical symptoms suggesting active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid is only required if there is a clinical suspicion of CNS involvement by leukemia during screening.
14. Subjects with immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
15. Subjects with a known medical history of progressive multifocal leukoencephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2023-01-18 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration(Cmax) | Measured on Day-3, Cyele1 Day1, Cycle1 Day15,Cycle2 Day1,Cycle3 Day1,Cycle4 Day1 (each cycle is 28 days)
Area under the plasma concentration versus time curve(AUC) | Measured on Day-3, Cyele1 Day1, Cycle1 Day15,Cycle2 Day1,Cycle3 Day1,Cycle4 Day1 (each cycle is 28 days)
The time to Cmax (Tmax) | Measured on Day-3, Cyele1 Day1, Cycle1 Day15,Cycle2 Day1,Cycle3 Day1,Cycle4 Day1 (each cycle is 28 days)
Half-life（t1/2） | Measured on Day-3, Cyele1 Day1, Cycle1 Day15,Cycle2 Day1,Cycle3 Day1,Cycle4 Day1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China